CLINICAL TRIAL: NCT05499143
Title: ImpACT for Developmental Coordination Disorder
Acronym: ImpactDCD
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0203
Record Dates: First submitted 2022-08-05; First posted 2022-08-12 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Developmental Coordination Disorder
Keywords: Child; Diagnostics; Early development; Neurodevelopmental disorders
MeSH Terms: conditions — Motor Skills Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of children with DCD or related movement difficulties
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — Online questionnaire impact for DCD - Belgian version

SUMMARY:
This study investigates the impact of Developmental Coordination Disorder on the child and its environment in Belgium within the following domains: diagnosis, activities and participation, school, therapy/support, and socio-emotional impact.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children living in Belgium
* Parents of children between 4 and 18 years old
* Parents of children who experience movement problems and/or there is a suspicion or diagnosis of DCD

Exclusion Criteria:

• Parents of children who have another other medical condition that would explain the movement difficulties (e.g. cerebral palsy, muscle disease,...)

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children who experience movement problems and/or there is a suspicion or diagnosis of DCD
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Impact of Developmental Coordination Disorder (DCD) | 1 year
  This translated and culturally adapted questionnaire will investigate the following domains: diagnosis, activities and participation, school, therapy/support, and socio-emotional impact.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Bar-On, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Licari MK, Alvares GA, Bernie C, Elliott C, Evans KL, McIntyre S, Pillar SV, Reynolds JE, Reid SL, Spittle AJ, Whitehouse AJO, Zwicker JG, Williams J. The unmet clinical needs of children with developmental coordination disorder. Pediatr Res. 2021 Oct;90(4):826-831. doi: 10.1038/s41390-021-01373-1. Epub 2021 Jan 27. PMID 33504966